CLINICAL TRIAL: NCT01952899
Title: Improvement of Care for ICU Patients With Delirium by Early Screening and Treatment
Brief Title: The ICU DElirium in Clinical PracTice Implementation Evaluation Study Screening and Treatment
Acronym: iDECePTIvE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Albert Schweitzer Hospital (Other); Ikazia Hospital, Rotterdam (Other); IJsselland Hospital (Unknown); Maasstad Hospital (Other); Sint Franciscus Gasthuis (Other)
Responsible Party: Principal Investigator, Z. Trogrlic, MSc / PhD-Student, Erasmus Medical Center
Other Study IDs: 80-82315-97-12025
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Delirium
Keywords: Intensive Care Unit; Delirium; Implementation; Guideline
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Albert Schweitzer Hospital
- Erasmus MC Academic Hospital
- Ikazia Hospital
- IJsselland Hospital
- Maasstad Hospital
- Sint Franciscus Gasthuis Hospital

SUMMARY:
Objective: Delirium is an important and frequently occurring complication in intensive care patients. However, screening and treatment of delirium is not in accordance with current national and international guidelines. The first objective of this prospective study is to describe the barriers and facilitators for guideline adherence. Second, investigators will develop a tailored implementation strategy. Finally, investigators will describe the effects of the tailored implementation on the adherence of the guideline in a pilot study. Design: Current practices, attitudes and deviations from a national (Dutch) delirium guideline will be assessed in a prospective before-measurement. Barriers and facilitators will be identified with surveys and focus group interviews. Adherence to the guideline will be studied in a before-after study in 7 ICUs in the Southwest of the Netherlands. Further, the effect of a multifaceted implementation strategy-guided implementation will be assessed with regard to important clinical outcomes, such as mortality and delirium incidence. Population: Professionals (Physicians/intensivists, nurses' and psychiatrists) and ICU patients. Intervention: The delirium guideline of the Netherlands Society of Intensive Care (NVIC) is implemented in this study. Implementation strategies: Barriers and facilitators will be determined in focus group interviews (n=7) with health care professionals resulting in a tailored guideline implementation strategy. In the development of the strategies specific attention will be paid to sustaining the guideline adherence. Main outcome: 1. Current practices; 2. Barriers and facilitators for guideline adherence; 3. Tailored implementation strategy; 4. Percentage of adherence to the guideline (early screening, prevention and treatment of delirium); 5. Effects of implementation on outcomes (economic, mortality, delirium incidence). Data analysis / power: The main effects, guideline adherence, will be evaluated by comparing the before and after measurements. Calculating from 90% power,2-sided alpha=0.01, 231 patients per periods will be sufficient to test the proposed adherence of 85%. Economic evaluation: The economic analysis will be performed from a health care perspective. Investigator will calculate and compare the direct medical costs of usual care (before) and care after implementation of the guideline. Additionally, the cost of the tailored guideline implementation process will be calculated. The economic analysis will be a cost-minimalization analysis.

ELIGIBILITY:
Inclusion Criteria:

* Screening delirium by all patients
* Measuring of guide line adherence for all professionals working on the ICU
* Implementation guideline: all professionals

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ICU patients and professionals
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-05 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Delirium guideline adherence | 36 monts
  1. Current practices;
  2. Barriers and facilitators for guideline adherence;
  3. Tailored implementation strategy;
  4. Percentage of adherence to the guideline (early screening, prevention and treatment of delirium);
  5. process evaluation in terms of relevant clinical outcomes, economic assessment, delirium incidence.
  6. Re-validation of delirium screening tools (CAM-ICU and ICDSC)

SECONDARY OUTCOMES:
Economic evaluation | 1 month
  The economic analysis will be performed from a health care perspective. Investigators will calculate and compare the direct medical costs of usual care (before) and care after implementation of the guideline. Additionally, the cost of the tailored guideline implementation process will be calculated. The economic analysis will be a cost-minimalization analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Erwin W. Ista, Dr, Study Director — Erasmus MC University Medical Center Rotterdam/ ZonMw; Mathieu van der Jagt, MD, PhD, Study Director — Department of Intensive Care, Erasmus MC - University Medical Center Rotterdam, Netherlands; Zoran Trogrlic, MSc, Principal Investigator — Department of Intensive Care, Erasmus MC - University Medical Center Rotterdam, Netherlands
Locations (1):
- Erasmus MC Academic Medica Center Rotterdam, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Smit L, Wiegers EJA, Trogrlic Z, Gommers D, Ista E, van der Jagt M. Risk factors for transitions and outcomes of subsyndromal delirium in the ICU: Post-hoc analysis of a prospective multicenter cohort study. J Crit Care. 2025 Aug;88:155041. doi: 10.1016/j.jcrc.2025.155041. Epub 2025 Mar 6. PMID 40054074
- [Derived] Smit L, Wiegers EJA, Trogrlic Z, Rietdijk WJR, Gommers D, Ista E, van der Jagt M. Prognostic significance of delirium subtypes in critically ill medical and surgical patients: a secondary analysis of a prospective multicenter study. J Intensive Care. 2022 Dec 20;10(1):54. doi: 10.1186/s40560-022-00644-1. PMID 36539913
- [Derived] Ista E, Trogrlic Z, Bakker J, Osse RJ, van Achterberg T, van der Jagt M. Improvement of care for ICU patients with delirium by early screening and treatment: study protocol of iDECePTIvE study. Implement Sci. 2014 Oct 2;9:143. doi: 10.1186/s13012-014-0143-7. PMID 25273854